CLINICAL TRIAL: NCT07079527
Title: Comparative Effects of Manual Positive End Expiratory Pressure and Non Invasive Continuous Air Pressure in COPD Patients
Brief Title: Effects of Manual Positive End Expiratory Pressure and Non-invasive Continuous Positive Air Pressure in COPD Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0357
Record Dates: First submitted 2025-07-03; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: COPD
Keywords: COPD, Posotive end expiratory pressure, CPAP
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Microcephaly, Primary Autosomal Recessive, 6 | interventions — Positive-Pressure Respiration; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual PEEP Therapy (Experimental): Participants in this group receive Manual Positive End Expiratory Pressure (PEEP) therapy. The therapy is administered using a tight-fitting mask that applies positive pressure at the end of expiration to keep alveoli open, enhance oxygenation, reduce airway collapse, and improve breathing efficiency. Sessions follow a standardized protocol over a 4-week period. All participants also receive Active Cycle of Breathing Techniques (ACBTs) as baseline therapy.
  Interventions: Device: Manual Positive End Expiratory Pressure (PEEP) Therapy
- Non-Invasive CPAP Therapy (Experimental): Participants in this group receive Non-Invasive Continuous Positive Airway Pressure (CPAP) therapy. CPAP delivers a constant level of positive pressure throughout the respiratory cycle using a non-invasive ventilator. This helps reduce the work of breathing, improve gas exchange, and relieve symptoms of dyspnea. The intervention is delivered according to a standardized protocol for 4 weeks, along with baseline ACBTs.
  Interventions: Device: Non-Invasive CPAP Therapy

INTERVENTIONS:
Device: Manual Positive End Expiratory Pressure (PEEP) Therapy — Participants in this group receive Manual Positive End Expiratory Pressure (PEEP) therapy. The intervention is delivered using a tight-fitting mask that applies positive pressure at the end of expiration, helping to keep the alveoli open, enhance oxygenation, and prevent airway collapse. The therapy is administered according to a structured protocol over a 4-week period, aiming to reduce breathlessness, improve lung function, and support ventilation. Along with PEEP, participants also receive baseline Active Cycle of Breathing Techniques (ACBTs) for airway clearance and breathing control.
  Arms: Manual PEEP Therapy
Device: Non-Invasive CPAP Therapy — Participants in this group receive Non-Invasive Continuous Positive Airway Pressure (CPAP) therapy. CPAP provides a constant level of positive pressure throughout the entire breathing cycle using a non-invasive ventilator and a full-face or nasal mask. This therapy improves gas exchange, reduces the work of breathing, and eases symptoms such as dyspnea. Like Group A, CPAP therapy is delivered following a standardized protocol for 4 weeks, and participants also perform baseline ACBTs to support respiratory function.
  Arms: Non-Invasive CPAP Therapy

SUMMARY:
This randomized clinical trial aims to compare the effectiveness of Manual Positive End Expiratory Pressure (PEEP) and Non-Invasive Continuous Positive Airway Pressure (CPAP) in patients with Chronic Obstructive Pulmonary Disease (COPD). A total of 42 patients will be randomly assigned to two groups: one receiving manual PEEP therapy and the other receiving CPAP therapy, over a 4-week period. The primary goal is to assess and compare improvements in respiratory rate, oxygen saturation (SpO₂), and patient-reported breathlessness and comfort using standardized tools such as pulse oximetry, digital spirometry, the Borg dyspnea scale, and the COPD Assessment Test. The study is designed as a single-blind randomized trial and will be conducted at Imran Idrees and Allama Iqbal Memorial Hospitals in Sialkot. The outcomes are expected to guide better non-invasive management strategies for COPD patients to enhance clinical outcomes and quality of life.

DETAILED DESCRIPTION:
This randomized clinical trial investigates the comparative effectiveness of Manual Positive End Expiratory Pressure (PEEP) and Non-Invasive Continuous Positive Airway Pressure (CPAP) in patients with Chronic Obstructive Pulmonary Disease (COPD). COPD is a progressive respiratory condition characterized by airflow limitation, leading to breathlessness, decreased exercise tolerance, and frequent hospitalizations. Non-invasive ventilation techniques such as PEEP and CPAP are widely used to manage respiratory symptoms and improve lung function in these patients, but direct comparisons of their efficacy remain limited.

A total of 42 patients with Stage 3 or 4 COPD, aged over 40 years, will be enrolled and randomly assigned to two groups:

Group A will receive manual PEEP therapy

Group B will receive non-invasive CPAP therapy

The intervention will last four weeks, and all patients will receive baseline treatment in the form of Active Cycle of Breathing Techniques (ACBTs). The study will be conducted at Imran Idrees Teaching Hospital and Allama Iqbal Memorial Hospital, Sialkot.

Primary outcome measures include improvements in:

Oxygen saturation (SpO₂)

Respiratory rate

Patient-reported breathlessness (using the Borg scale)

Quality of life and symptom severity (using the COPD Assessment Test)

Data collection tools include pulse oximetry, digital spirometry (for FEV₁, FVC, PEF), and standardized questionnaires. The study uses a single-blind design, where the assessor is blinded to the group allocation.

The purpose is to determine which intervention-manual PEEP or CPAP-offers superior clinical outcomes, patient comfort, and symptom relief. Findings from this research aim to support evidence-based decision-making for non-invasive COPD management in clinical settings.

ELIGIBILITY:
Inclusion Criteria:

* Age>40years old
* SevereCOPDpatients with Stage 3 & 4 according to Gold Criteria
* Notcurrently experiencing an acute exacerbation.
* Baseline Forced Expiratory Volume in 1 second (FEV1) < 70% of predicted
* Ability to provide informed consent.

Exclusion Criteria:

* Othersignificant respiratory diseases (e.g., asthma, pulmonary fibrosis, cystic fibrosis)
* Invasive mechanical ventilation
* Pregnant or Breastfeeding women
* Cardiac arrhythmias or instability

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-07-28 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Change in SpO₂ (Oxygen Saturation) from Baseline to Post-Intervention | 4 weeks
  Oxygen saturation (%) will be measured using a pulse oximeter before and after the 4-week intervention. The average change in SpO₂ will be compared within and between both groups.
Change in Respiratory Rate (RR) from Baseline to Post-Intervention | 4 weeks
  Respiratory rate (breaths per minute) will be recorded at baseline and after 4 weeks. Lower respiratory rate post-intervention reflects clinical improvement.
Borg Dyspnea Scale Score from Baseline to Post-Intervention at 4 weeks | 4 weeks
  The Borg Dyspnea Scale, a 0-10 point subjective scale, will be used to evaluate the severity of dyspnea in COPD patients. A score of 0 represents no breathlessness, and a score of 10 represents maximal breathlessness. Higher scores indicate worse outcomes (i.e., more severe dyspnea). Measurements will be taken at baseline and after the 8-week intervention. The primary analysis will focus on the change in median score from pre- to post-intervention within and between groups.
  MaximumHigher scores indicate worse dyspnea (more severe breathlessness) score: 10

SECONDARY OUTCOMES:
Change in Distance Walked during 6-Minute Walk Test (6MWT) | 4 weeks
  Total distance walked (in meters) during the 6MWT will be recorded. Higher distance reflects improved functional capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Arjumand Bano, Ms CPPT, Principal Investigator — Riphah International University
Locations (1):
- Arjumand, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No